CLINICAL TRIAL: NCT03297632
Title: Functionally Designed Resistance Exercise With the Aim of Improving Balance, Muscle Strength, Muscle Mass and Physical Function of the Elderly: a Randomized Controlled Study
Brief Title: Improving Muscle Strength, Mass and Physical Function in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Region Västerbotten (Other Government)
Responsible Party: Principal Investigator, Anna Nordström, Adjunct Professor, Region Västerbotten
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VCC-LIFE-3
Record Dates: First submitted 2017-09-18; First posted 2017-09-29 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Muscle Weakness; Fall; Sarcopenia
MeSH Terms: conditions — Muscle Weakness; Sarcopenia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (Experimental): Receives instructor-based functional resistance exercise. 45 minutes per session. 3 times per week, during 10 weeks in total.
  Interventions: Behavioral: Functional resistance exercise
- Control group (No Intervention): Asked to normally active according to their current lifestyle
- Home-based group (Active Comparator): Receives home-based exercises with written instructions and digital video support. 45 minutes per session. 3 times per week, during 10 weeks in total.
  Interventions: Behavioral: Functional resistance exercise

INTERVENTIONS:
Behavioral: Functional resistance exercise — Functional resistance program designed for older individuals with low muscle mass and muscle strength. The goal is to implement exercises that are possible for the participants to also perform in their home environment, through the use of basic equipment.
  Arms: Home-based group; Intervention Group

SUMMARY:
Falls and fractures are serious and costly events for elderly individuals: they cause functional impairments, increase mortality and contribute to huge healthcare costs for the society. The number of falls, and following consequences, are expected to increase in society as the proportion of the elderly population will increase, therefore it is crucial to be able to detect and prevent falls and fractures in the population. The investigators have previously published results that objective measurements of postural balance can predict fall risk in 70-year-olds in Umeå and subsequently investigated whether balance can be improved through 4-week balance exercise program. However, preliminary results suggest that the frequency and duration of exercise should be longer than 3 times a week for 4 weeks to produce effects. Furthermore, there is also evidence indicating a link between muscle weakness and fall risk in elderly subjects, while research findings show that it is possible for older individuals to influence muscle strength and muscle mass with resistance exercise. Functional strength training can also positively influence the balance. In this context, the investigators aim to investigate whether a 10-week resistance exercise program may positively affect balance, muscle strength, muscle mass and physical function, with the aim of preventing future falls and fractures in the population.

DETAILED DESCRIPTION:
Background:

Falls and fall-related injuries are major health concerns for elderly individuals; they cause functional decline and increased mortality, as well as incurring vast health care costs for society. Occurrences and consequences of falls are expected to increase globally with the growing number of elderly individuals. Hence, the improved detection of potential fall risk markers is of importance when predicting individuals at risk for falls and subsequently for improving strategies in fall-prevention. Falling can be the end result of intrinsic and extrinsic factors negatively affecting an individual's ability to maintain balance, which are often revealed during sequences of body movement. Balance can be both dynamically and statically measured, the latter involves having the individual in a stationary standing position, from which results researchers have proposed impaired postural stability as a risk factor for falling. However, evidence regarding the association of postural instability with prospective falls is limited, and population-based cohort studies in this field are scarce. Other shortcomings of previous studies include the use of retrospective study designs, which increase the risks of recall bias and the identification of risk factors as the result of falls.

Postural instability is preferably investigated using objective measures of posturography, which has advantages over regular clinical assessments since it reduces test performance variability and avoids the subjective nature of scoring systems. Recently, researchers has analyzed the performance of the Wii Balance Board (WBB) as an instrument for measuring postural instability, revealing excellent concurrent validity and an ability to complement existing fall assessments. However, these findings needed to be evaluated in a population-based sample with a rich set of covariates. Hence, the investigators performed a prospectively observational study to investigate how objective measures of postural sway predicted prospective falls in a cohort of more than 1800 community-dwelling men and women, all of whom were 70 years of age at the time of the investigation.

The results revealed that impaired postural stability can increase the risk of incident falls by 75 to 90% among older adults in the highest quintile of postural sway, measured during trials of both eyes open and eyes closed. One of the conclusions was that it would be valuable to examine the clinical utility of the investigated parameters in future studies, compare performance to established clinical balance tests, and to investigate whether strategies to improve balance would reduce the fall risk. Thus, in a follow-up study the investigators examined wether they could reduce the increased postural sway of participants who was identified as having abnormal balance values, based on previous measurements. The investigators also examined participants' functional balance through Time-Up-and-GO (TUG) performance, together with measures of muscle strength and validated questionnaires on Fear of Falling and Falls Efficacy. This follow-up study was conducted as a randomized intervention study, with a total of 52 individuals recruited from the existing HAI study cohort, with measures of postural sway in the 5th quintile, which indicated impaired balance function. The intervention group performed three supervised group training sessions a week, consisting of 30 minutes of balance training for 4 weeks while the control group received a health consultation highlighting the importance of physical activity and balance exercise. Preliminary data indicated that the exercise intervention had little to no effect on selected measures on balance, strength and physical function. Thus, it may seem that a exercise volume of 4 weeks of progressive balance exercise, 3 sessions per week, might be to low to produce beneficial effects.

The results from this previous study indicated the need for a more comprehensive exercise program in order to produce beneficial effects on balance, strength and physical function, and in the long term, fall prevention. Previous research has shown that low muscle strength together with low muscle mass, also known as sarcopenia, independently predicts falls, fractures and overall poor health. However, a growing body of evidence also indicates that older individuals are able to counteract the trend of age-related loss of muscle mass, as well as improve dynamic balance, through the use of resistance exercise. For older individuals, it is recommended that the exercise regimen lasts for 10-12 weeks, with 3 exercise sessions each week, in order to produce effects on muscle strength, muscle mass and physical function, which is a higher total exercise volume than what was used in the balance exercise study.

Aims:

1. The primary aim of the current study is to investigate the effect and feasibility of a 10-week instructor-supervised resistance exercise program designed for older individuals with low muscle mass. The goal is to implement exercises that are possible for the participants to also perform in their home environment, through the use of basic equipment.
2. A secondary aim is to evaluate the effect of the very same exercise program, recorded in digital videos and written instructions, to be used by the participant in their own residence or similar location.

Methods:

Recruitment is based on participants previously enrolled in the Healthy Ageing Initiative (HAI) health examination, an on-going population based cohort study which invites all 70-year-olds in the Umeå municipality to participate. Eligible participants for this study will be drawn from the lowest quintile of muscle mass (pre-sarcopenia) for men and women, based on Dual-Energy X-ray Absorptiometry (DEXA, GE Healthcare, Lunar, Madison, WI, USA) measurements in the HAI study and criteria taken from the European definition on sarcopenia. Participants are first contacted by telephone where they receive information about the study and are invited to participate. Upon agreement, participants are randomized either to the control group, a home-based training group or instructor-led training group. The latter group is offered instructor-based weight training in groups, three times a week for 10 weeks. The exercise program is designed to engage whole-body muscle groups, with focus on leg and core musculature, as well as being functional and include movements and muscle actions important for active daily living. The home-based training includes 10 weeks of the same exercise program, performed at home with digital support. The control group are offered access to training instructions as well as digital support during follow up 6 months after the start of the study. In addition, all participants receive cost-free training equipment for home use.

Testing is performed at baseline, after the intervention period during follow-up at 10 weeks, as well as 6 months after baseline. The following tests and outcomes are included:

1. Primary outcome is Short Physical Performance Battery (SPPB) test score. The SPPB includes several functional tests evaluating leg strength and power, postural stability and gait speed. The SPPB is a common and validated clinical test of physical function.
2. Secondary outcomes include:

   * Objective measurement of postural stability, using the Wii Balance Board (WBB; Nintendo, Kyoto, Japan) device, described and validated in a previously published study (8). Each participant conducts two 60-s trials in a quiet stance, consisting of eyes-open (EO) and eyes-closed (EC) conditions. Participants are instructed to maintain an upright position throughout the test, stand relaxed and avoid any arm or head movement. The WBB measures total centre of pressure (COP) sway length, representing the sum of postural sway in the anteroposterior and mediolateral directions.
   * Isometric muscle strength, tested by using a hydraulic hand dynamometer (Jamar; Patterson Medical, Warrenville, IL, USA) to measure each participant's maximum grip strength in the non-dominant hand. Participants are instructed to keep the arm at a 90° angle and to maintain the elbow in proximity to the waist during the test. The maximum value obtained in two consecutive attempts is recorded.
   * Appendicular lean mass (ALM), measured with a iDXA device (GE Healthcare, Lunar, Madison, WI, USA). Measurements are based on whole-body scans with a duration of approximately 8 minutes. An ALM index is subsequently calculated by combining the total muscle mass in arms and legs and dividing by height squared (ALM/m2) of the participant, according to the standards set by the European Working Group on Sarcopenia in Older People (EWGSOP).
   * Timed-Up-and-Go (TUG) test performance, a test commonly used by clinicians to assess lower leg muscle strength, gait performance, and overall functional mobility in elderly individuals. In this test, each participant are asked to rise unaided from an armchair and walk forward 3 meters until he or she reached a line marked on the floor, then to turn around and return to a seated position in the chair. Test leaders provide instructions and measure total testing time using a stopwatch.
   * Objective measures of physical activity, measured by triaxial accelerometers (GT3X., 4.6 3.3 1.5 cm; Actigraph, Pensacola, FL) for 7 days. These devices are capable of measuring acceleration in the range of 6 G. Measured accelerations are digitalized, transformed into "counts," and stored in a resilient flash memory. Participants wear the accelerometers on their non-dominant hips, removing them only when showering, swimming, or during nighttime sleep. They also receive instructions to be normally active during the measurement period, to obtain accurate reflections of their lifestyles.
   * Fear of Falling, using the validated Falls Efficacy Scale-International (FES-I) questionnaire.
   * Self-recalled physical activity, using the validated International Physical Activity Questionnaire (IPAQ) Furthermore, the investigators aim to investigate postural stability, TUG test performance, Fear of Falling and self-recalled physical activity 4 weeks after baseline, in order to facilitate comparison between resistance exercise to the balance exercise program performed in the previous 4- week randomized controlled trial (Ethical approval Dnr: 2017-132-31).

Statistical power analysis:

The power calculation is based on the main outcome for the study, i.e. the short physical performance battery (SPPB). SPPB was previously tested in 2.710 older sample of Italian adults with a mean age of 75 (range 65-97). Women scored 7.79±3.22 (mean ± standard deviation) and men scored 9.03±3.12. In the present study the investigators will include a more homogeneous sample of younger age but with pre-sarcopenia. Therefore, estimations are that the score in this sample at baseline will be 8±2.5. From a previous study including 424 elderly persons at risk for disability (ages 70-89 years), it was shown that SPPB increased 16% from 6 months of moderate physical activity in the intervention group, which decreased slightly to 13.3% after 1 year. These effects were significantly different compared to in the control group (p<0.001), where no changes were seen in SPPB. There was slightly better effect of training in women and those with a SPPB of at least 7 at baseline. Based on these figures the investigators estimate that the intervention group will increase 12% in SPPB during the 10 weeks of training, with no changes in the control group. Based on these assumptions, 107 persons will be needed in each group, to have 80% power to detect a two-sided effect with α-level of 0.05.

In the first round of enrollment starting this fall, the investigators have begun randomizing 36 participants to each group. The aim is to continue and enroll remaining participants during the second round starting late spring/early fall 2018.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the Healthy Ageing Initiative (HAI) study
* Appendicular lean mass index in the lowest 20% measured with the iDXA in the HAI study, separate for men and women.

Exclusion Criteria:

* Unable to be present during all 10 weeks of exercise.

Ages: 70 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2017-09-04 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Postural Stability performance | Change in Postural Stability performance at 10 and 34 weeks
  Postural stability measurement task from the Short Physical Performance Battery (SPPB), containing bipedal, semi-tandem and tandem stances. Measured in seconds, up to a maximal value of 10 seconds.
Change in Gait Speed | Change in Gait Speed at 10 and 34 weeks
  Gait speed measurement task from the Short Physical Performance Battery (SPPB). Measured in the seconds it takes to walk 4 meters.
Change in Chair Stand performance | Change in Chair stand performance at 10 and 34 weeks
  Chair stand measurement task from the Short Physical Performance Battery (SPPB). Measures in the time it takes to stand up 5 times.

SECONDARY OUTCOMES:
Change in Postural Sway | Change in Baseline Postural Sway at 10 and 34 weeks
  Total postural sway length, measured objectively during trials of eyes open and eyes closed, during 60 seconds each
Change in Isometric Muscle Strength | Change in Baseline Isometric Muscle Strength at 10 and 34 weeks
  Measured by using a hydraulic hand dynamometer. The maximum value obtained in two consecutive attempts is recorded.
Change in Appendicular Muscle Mass | Change in Baseline Appendicular Muscle Mass at 10 and 34 weeks
  Measured with a iDXA device. Measurements are based on whole-body scans with a duration of approximately 8 minutes.
Change in TUG test performance | Change in Baseline TUG test performance at 10 and 34 weeks
  The Timed-Up-and-Go test is commonly used by clinicians to assess lower leg muscle strength, gait performance, and overall functional mobility in elderly individuals
Change in Physical Activity | Change in Baseline Physical Activity at 10 and 34 weeks
  Objective measures through the use of triaxial accelerometers
Change in Fear of Falling | Change in Baseline Fear of Falling at 10 and 34 weeks
  Assessed with the validated Falls Efficacy Scale-International questionnaire
Change in self-recalled Physical Activity | Change in Baseline self-recalled Physical Activity at 10 and 34 weeks
  Assessed with the validated International Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Livsmedicin (LIFE), Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stel VS, Smit JH, Pluijm SM, Lips P. Consequences of falling in older men and women and risk factors for health service use and functional decline. Age Ageing. 2004 Jan;33(1):58-65. doi: 10.1093/ageing/afh028. PMID 14695865
- [Background] Wolinsky FD, Fitzgerald JF, Stump TE. The effect of hip fracture on mortality, hospitalization, and functional status: a prospective study. Am J Public Health. 1997 Mar;87(3):398-403. doi: 10.2105/ajph.87.3.398. PMID 9096540
- [Background] Rizzo JA, Friedkin R, Williams CS, Nabors J, Acampora D, Tinetti ME. Health care utilization and costs in a Medicare population by fall status. Med Care. 1998 Aug;36(8):1174-88. doi: 10.1097/00005650-199808000-00006. PMID 9708590
- [Background] Masud T, Morris RO. Epidemiology of falls. Age Ageing. 2001 Nov;30 Suppl 4:3-7. doi: 10.1093/ageing/30.suppl_4.3. No abstract available. PMID 11769786
- [Background] Robinovitch SN, Feldman F, Yang Y, Schonnop R, Leung PM, Sarraf T, Sims-Gould J, Loughin M. Video capture of the circumstances of falls in elderly people residing in long-term care: an observational study. Lancet. 2013 Jan 5;381(9860):47-54. doi: 10.1016/S0140-6736(12)61263-X. Epub 2012 Oct 17. PMID 23083889
- [Background] Tinetti ME, Speechley M, Ginter SF. Risk factors for falls among elderly persons living in the community. N Engl J Med. 1988 Dec 29;319(26):1701-7. doi: 10.1056/NEJM198812293192604. PMID 3205267
- [Background] Maki BE, Holliday PJ, Topper AK. A prospective study of postural balance and risk of falling in an ambulatory and independent elderly population. J Gerontol. 1994 Mar;49(2):M72-84. doi: 10.1093/geronj/49.2.m72. PMID 8126355
- [Background] Piirtola M, Era P. Force platform measurements as predictors of falls among older people - a review. Gerontology. 2006;52(1):1-16. doi: 10.1159/000089820. PMID 16439819
- [Background] Lord SR, Sambrook PN, Gilbert C, Kelly PJ, Nguyen T, Webster IW, Eisman JA. Postural stability, falls and fractures in the elderly: results from the Dubbo Osteoporosis Epidemiology Study. Med J Aust. 1994 Jun 6;160(11):684-5, 688-91. PMID 8202002
- [Background] Moe-Nilssen R, Nordin E, Lundin-Olsson L; Work Package 3 of European Community Research Network Prevention of Falls Network Europe. Criteria for evaluation of measurement properties of clinical balance measures for use in fall prevention studies. J Eval Clin Pract. 2008 Apr;14(2):236-40. doi: 10.1111/j.1365-2753.2007.00839.x. PMID 18324932
- [Background] Howcroft J, Kofman J, Lemaire ED. Review of fall risk assessment in geriatric populations using inertial sensors. J Neuroeng Rehabil. 2013 Aug 8;10(1):91. doi: 10.1186/1743-0003-10-91. PMID 23927446
- [Background] Visser JE, Carpenter MG, van der Kooij H, Bloem BR. The clinical utility of posturography. Clin Neurophysiol. 2008 Nov;119(11):2424-36. doi: 10.1016/j.clinph.2008.07.220. Epub 2008 Sep 12. PMID 18789756
- [Background] Scaglioni-Solano P, Aragon-Vargas LF. Validity and reliability of the Nintendo Wii Balance Board to assess standing balance and sensory integration in highly functional older adults. Int J Rehabil Res. 2014 Jun;37(2):138-43. doi: 10.1097/MRR.0000000000000046. PMID 24445863
- [Background] Kwok BC, Clark RA, Pua YH. Novel use of the Wii Balance Board to prospectively predict falls in community-dwelling older adults. Clin Biomech (Bristol). 2015 Jun;30(5):481-4. doi: 10.1016/j.clinbiomech.2015.03.006. Epub 2015 Mar 11. PMID 25796535
- [Background] Johansson J, Nordstrom A, Gustafson Y, Westling G, Nordstrom P. Increased postural sway during quiet stance as a risk factor for prospective falls in community-dwelling elderly individuals. Age Ageing. 2017 Nov 1;46(6):964-970. doi: 10.1093/ageing/afx083. PMID 28531243
- [Background] Cederholm T, Cruz-Jentoft AJ, Maggi S. Sarcopenia and fragility fractures. Eur J Phys Rehabil Med. 2013 Feb;49(1):111-7. PMID 23575205
- [Background] Borde R, Hortobagyi T, Granacher U. Dose-Response Relationships of Resistance Training in Healthy Old Adults: A Systematic Review and Meta-Analysis. Sports Med. 2015 Dec;45(12):1693-720. doi: 10.1007/s40279-015-0385-9. PMID 26420238
- [Background] Yu W, An C, Kang H. Effects of Resistance Exercise Using Thera-band on Balance of Elderly Adults: A Randomized Controlled Trial. J Phys Ther Sci. 2013 Nov;25(11):1471-3. doi: 10.1589/jpts.25.1471. Epub 2013 Dec 11. PMID 24396213
- [Background] de Labra C, Guimaraes-Pinheiro C, Maseda A, Lorenzo T, Millan-Calenti JC. Effects of physical exercise interventions in frail older adults: a systematic review of randomized controlled trials. BMC Geriatr. 2015 Dec 2;15:154. doi: 10.1186/s12877-015-0155-4. PMID 26626157
- [Background] Iolascon G, Di Pietro G, Gimigliano F, Mauro GL, Moretti A, Giamattei MT, Ortolani S, Tarantino U, Brandi ML. Physical exercise and sarcopenia in older people: position paper of the Italian Society of Orthopaedics and Medicine (OrtoMed). Clin Cases Miner Bone Metab. 2014 Sep;11(3):215-21. PMID 25568656
- [Background] Veronese N, Bolzetta F, Toffanello ED, Zambon S, De Rui M, Perissinotto E, Coin A, Corti MC, Baggio G, Crepaldi G, Sergi G, Manzato E. Association between Short Physical Performance Battery and falls in older people: the Progetto Veneto Anziani Study. Rejuvenation Res. 2014 Jun;17(3):276-84. doi: 10.1089/rej.2013.1491. Epub 2014 Jun 11. PMID 24387140
- [Background] LIFE Study Investigators; Pahor M, Blair SN, Espeland M, Fielding R, Gill TM, Guralnik JM, Hadley EC, King AC, Kritchevsky SB, Maraldi C, Miller ME, Newman AB, Rejeski WJ, Romashkan S, Studenski S. Effects of a physical activity intervention on measures of physical performance: Results of the lifestyle interventions and independence for Elders Pilot (LIFE-P) study. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1157-65. doi: 10.1093/gerona/61.11.1157. PMID 17167156
- [Derived] Vikberg S, Sorlen N, Branden L, Johansson J, Nordstrom A, Hult A, Nordstrom P. Effects of Resistance Training on Functional Strength and Muscle Mass in 70-Year-Old Individuals With Pre-sarcopenia: A Randomized Controlled Trial. J Am Med Dir Assoc. 2019 Jan;20(1):28-34. doi: 10.1016/j.jamda.2018.09.011. Epub 2018 Nov 7. PMID 30414822